CLINICAL TRIAL: NCT01469234
Title: A Double-Blind, Parallel, Randomized, Placebo Controlled Trial to Evaluate Onset of Action of Loratadine and Fexofenadine in Subjects With Seasonal Allergic Rhinitis in a Pollen Challenge Chamber
Brief Title: A Study of Onset of Action of Loratadine and Fexofenadine in Participants With Seasonal Allergic Rhinitis (P08712)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18126; PT11-37 (Other: Consumer Health Care); P08712 (Other: Merck)
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — Loratadine; fexofenadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- loratadine (Experimental): Participants will receive one dose of loratadine following randomization at 120 minutes of exposure during visit 4.
  Interventions: Drug: loratadine; Drug: placebo to fexofenadine
- fexofenadine (Experimental): Participants will receive one dose of fexofenadine following randomization at 120 minutes of exposure during visit 4.
  Interventions: Drug: fexofenadine; Drug: placebo to loratadine
- placebo (Placebo Comparator): Participants will receive one dose of placebo following randomization at 120 minutes of exposure during visit 4.
  Interventions: Drug: placebo to loratadine; Drug: placebo to fexofenadine

INTERVENTIONS:
Drug: loratadine — loratadine, one 10 mg tablet, orally
  Other Names: SCH 029851
  Arms: loratadine
Drug: fexofenadine — fexofenadine, one 180 mg tablet, orally
  Arms: fexofenadine
Drug: placebo to loratadine — one tablet, orally
  Arms: fexofenadine; placebo
Drug: placebo to fexofenadine — one tablet, orally
  Arms: loratadine; placebo

SUMMARY:
The purpose of this study is to determine the onset of action of two commercially available over-the-counter antihistamines (Loratadine and

Fexofenadine) in a model of seasonal allergic rhinitis (SAR). Participants undergo sensitization exposures to Mountain Cedar (juniperus ashei) pollen in a Biogenics Research Chamber; those who demonstrate an adequate allergic response determined by the Major Symptom Complex (MSC) score will then receive drug.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of child bearing potential must demonstrate a negative

urine pregnancy test at Screening (Visit 1) and Visit 4 (prior to randomization) and agree to use (and/or have their partner use) 2 acceptable methods of birth control beginning at the Screening visit and throughout the study.

* Willing to stop use of current decongestant and allergy medications at the start of the washout period (Visit 1) and during the trial.
* Documented history or participant-reported history of seasonal allergic rhinitis caused by mountain cedar pollen within the last 2 years and documented or participant-reported symptoms over at least the last 2 mountain cedar allergy seasons.
* Documented skin testing (prick with wheal ≥ 4 mm larger than the diluent) within the last 1 year to mountain cedar pollen present.
* Capable of reading English.
* Body mass index (BMI) <35.

Exclusion Criteria:

* Any significant medical condition which, in the judgment of the investigator, is a contraindication to the use of loratadine, fexofenadine or might interfere with the trial. These may include thyroid disease (e.g., hyperthyroidism, hypothyroidism), uncontrolled diabetes mellitus, coronary heart disease, ischemic heart disease, elevated intraocular pressure, prostatic hypertrophy.
* Have started allergen immunotherapy within 1 month preceding enrollment or participants starting allergen immunotherapy or anticipating immunotherapy dose change during the trial. Xolair (omalizumab) may not be used within 4 years prior to trial participation.
* Known allergy or intolerance to loratadine, desloratadine, or fexofenadine.
* History of rhinitis medicamentosa.
* Use of systemic (oral, rectal, injectable), topical (up to 1% topical hydrocortisone is permitted), or nasal corticosteroids in the last 30 days or current or expected use of disallowed medications as listed in the protocol.
* Asthma, with the exception of mild intermittent asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Loratadine: Participants received one dose of loratadine following randomization at 120 minutes of exposure during visit 4.
- Fexofenadine: Participants received one dose of fexofenadine following randomization at 120 minutes of exposure during visit 4.
- Placebo: Participants received one dose of placebo following randomization at 120 minutes of exposure during visit 4.
Period: Overall Study
Arm/Group | Loratadine | Fexofenadine | Placebo
Started | 85 | 85 | 85
Completed | 85 | 85 | 85
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loratadine | Fexofenadine | Placebo | Total
Number analyzed (Participants) | 85 | 85 | 85 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (13.52) | 43.1 (12.21) | 40.6 (12.56) | 41.7 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 53 | 53 | 157
  Male | 34 | 32 | 32 | 98

OUTCOME MEASURES:

1. Primary Outcome: Mean Major Symptom Complex (MSC) Score by Post-Treatment Evaluation Time Point (From 180 Minutes to 300 Minutes)
Description: The MSC Score is calculated as the sum of 5 individual symptom scores for Runny Nose, Itchy Nose, Sneezing, Watery Eyes, and Itchy Eyes. Each individual symptom is rated on a 5-point scale of severity: 0 = None (No symptoms), 1 = MILD (Symptom is present, but easily tolerated), 2 = MODERATE (Awareness of symptoms, bothersome, but tolerable), 3 = SEVERE (Definite awareness of symptoms, difficult to tolerate but does not interfere with activities), 4 = VERY SEVERE (Difficult to tolerate and interferes with the activities of daily living). The total MSC score ranges from 0 - 25. Increasing scores are associated with increasing severity.
Time Frame: From time of sensitization (time 0) to end of visit (~8 hours)
Population: Participants in the Intent-to-Treat (ITT) Population (defined as all participants who successfully exhibited appropriate sensitivity and were randomized to study treatment) who had data available.
  N=Number of Participants Analyzed, n=number of participants with data available at the given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Loratadine | Fexofenadine | Placebo
Number analyzed (Participants) | 85 | 85 | 85
units on a scale
  180 minutes (n=85, n=85, n=85) | 7.4 (4.51) | 6.7 (4.86) | 8.5 (5.07)
  195 minutes (n=85, n=85, n=85) | 7.5 (4.84) | 6.7 (4.87) | 8.9 (5.31)
  210 minutes (n=85, n=85, n=85) | 7.3 (4.73) | 6.5 (4.87) | 8.7 (5.28)
  225 minutes (n=85, n=85, n=85) | 7.4 (4.63) | 6.5 (4.70) | 8.5 (5.36)
  240 minutes (n=84, n=85, n=85) | 7.4 (4.76) | 6.5 (4.43) | 8.3 (5.38)
  255 minutes (n=85, n=85, n=85) | 7.1 (4.78) | 6.3 (4.47) | 8.4 (5.51)
  270 minutes (n=85, n=85, n=85) | 7.0 (4.67) | 6.4 (4.50) | 8.4 (5.56)
  285 minutes (n=85, n=85, n=85) | 7.3 (4.52) | 6.9 (4.76) | 8.7 (5.76)
  300 minutes (n=84, n=85, n=85) | 7.1 (4.54) | 6.5 (4.65) | 8.4 (5.58)

2. Secondary Outcome: Mean Individual Symptom Score for Runny Nose by Post-Treatment Evaluation Time Point
Description: The individual symptom score for Runny Nose was rated on a 5-point
  scale of severity using the following scale: 0 = None (No symptoms), 1 = MILD (Symptom is present, but easily tolerated), 2 = MODERATE (Awareness of symptoms, bothersome, but tolerable), 3 = SEVERE (Definite awareness of symptoms, difficult to tolerate but does not interfere with activities), 4 = VERY SEVERE (Difficult to tolerate and interferes with the activities of daily living). The Runny Nose symptom score ranges from 0 - 5. Increasing scores are associated with increasing severity.
Time Frame: From time of sensitization (time 0) to end of visit (~8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Loratadine | Fexofenadine | Placebo
Number analyzed (Participants) | 85 | 85 | 85
units on a scale
  0 minutes | 3.4 (0.77) | 3.2 (0.78) | 3.3 (0.89)
  15 minutes | 3.1 (0.85) | 3.0 (0.91) | 3.0 (1.09)
  30 minutes | 3.0 (0.95) | 2.9 (0.99) | 2.9 (1.14)
  45 minutes | 2.8 (0.99) | 2.6 (1.05) | 2.8 (1.15)
  60 minutes | 2.7 (1.06) | 2.3 (1.02) | 2.7 (1.20)
  75 minutes | 2.6 (1.06) | 2.2 (1.08) | 2.6 (1.20)
  90 minutes | 2.4 (1.04) | 2.1 (1.08) | 2.4 (1.28)
  105 minutes | 2.4 (1.10) | 2.1 (1.03) | 2.5 (1.16)
  120 minutes | 2.1 (1.07) | 2.0 (1.00) | 2.3 (1.18)
  135 minutes | 2.2 (1.12) | 2.0 (1.07) | 2.4 (1.19)
  150 minutes | 2.3 (1.10) | 2.0 (1.07) | 2.4 (1.20)
  165 minutes | 2.2 (1.07) | 1.8 (1.14) | 2.3 (1.18)
  180 minutes | 2.1 (1.20) | 1.9 (1.20) | 2.3 (1.17)
  195 minutes | 2.1 (1.27) | 1.9 (1.21) | 2.4 (1.20)
  210 minutes | 2.0 (1.23) | 1.8 (1.22) | 2.3 (1.24)
  225 minutes | 2.1 (1.22) | 1.8 (1.24) | 2.3 (1.19)
  240 minutes | 2.0 (1.23) | 1.8 (1.19) | 2.2 (1.20)
  255 minutes | 2.0 (1.30) | 1.7 (1.15) | 2.3 (1.28)
  270 minutes | 1.9 (1.30) | 1.8 (1.10) | 2.3 (1.35)
  285 minutes | 2.1 (1.24) | 1.9 (1.15) | 2.3 (1.31)
  300 minutes | 2.0 (1.26) | 1.8 (1.14) | 2.3 (1.28)
  315 minutes | 2.1 (1.25) | 1.8 (1.17) | 2.4 (1.30)
  330 minutes | 2.2 (1.26) | 1.8 (1.18) | 2.3 (1.31)
  345 minutes | 2.1 (1.27) | 1.8 (1.17) | 2.4 (1.32)
  360 minutes | 2.1 (1.29) | 1.9 (1.23) | 2.3 (1.33)

3. Secondary Outcome: Mean Individual Symptom Score for Itchy Nose by Post-Treatment Evaluation Time Point
Description: The individual symptom score for Itchy Nose was rated on a 5-point
  scale of severity using the following scale: 0 = None (No symptoms), 1 = MILD (Symptom is present, but easily tolerated), 2 = MODERATE (Awareness of symptoms, bothersome, but tolerable), 3 = SEVERE (Definite awareness of symptoms, difficult to tolerate but does not interfere with activities), 4 = VERY SEVERE (Difficult to tolerate and interferes with the activities of daily living). The Itchy Nose symptom score ranges from 0 - 5. Increasing scores are associated with increasing severity.
Time Frame: From time of sensitization (time 0) to end of visit (~8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Loratadine | Fexofenadine | Placebo
Number analyzed (Participants) | 85 | 85 | 85
units on a scale
  0 minutes | 3.3 (0.74) | 3.3 (0.73) | 3.4 (0.77)
  15 minutes | 3.1 (0.84) | 3.2 (0.81) | 3.1 (0.93)
  30 minutes | 2.8 (0.97) | 2.8 (0.97) | 2.8 (0.99)
  45 minutes | 2.7 (1.02) | 2.6 (0.96) | 2.8 (1.04)
  60 minutes | 2.6 (1.09) | 2.4 (1.05) | 2.6 (1.07)
  75 minutes | 2.4 (1.16) | 2.3 (1.14) | 2.5 (1.19)
  90 minutes | 2.3 (1.10) | 2.1 (1.07) | 2.4 (1.17)
  105 minutes | 2.2 (1.08) | 2.1 (1.10) | 2.4 (1.10)
  120 minutes | 1.9 (1.14) | 1.8 (1.12) | 2.1 (1.20)
  135 minutes | 2.0 (1.12) | 1.8 (1.17) | 2.2 (1.22)
  150 minutes | 2.1 (1.06) | 1.8 (1.19) | 2.2 (1.18)
  165 minutes | 2.0 (1.09) | 1.7 (1.22) | 2.2 (1.14)
  180 minutes | 2.0 (1.16) | 1.8 (1.25) | 2.2 (1.12)
  195 minutes | 1.9 (1.23) | 1.7 (1.22) | 2.2 (1.20)
  210 minutes | 2.0 (1.25) | 1.7 (1.28) | 2.2 (1.20)
  225 minutes | 1.9 (1.18) | 1.7 (1.27) | 2.2 (1.25)
  240 minutes | 1.9 (1.14) | 1.7 (1.24) | 2.2 (1.24)
  255 minutes | 1.8 (1.24) | 1.7 (1.21) | 2.2 (1.30)
  270 minutes | 1.9 (1.18) | 1.7 (1.25) | 2.1 (1.31)
  285 minutes | 1.9 (1.17) | 1.8 (1.22) | 2.2 (1.29)
  300 minutes | 1.8 (1.19) | 1.8 (1.20) | 2.1 (1.32)
  315 minutes | 1.8 (1.26) | 1.8 (1.22) | 2.2 (1.38)
  330 minutes | 1.8 (1.16) | 1.7 (1.25) | 2.1 (1.31)
  345 minutes | 1.9 (1.23) | 1.7 (1.29) | 2.2 (1.36)
  360 minutes | 1.8 (1.22) | 1.8 (1.32) | 2.2 (1.38)

4. Secondary Outcome: Mean Individual Symptom Scores for Sneezing by Post-Treatment Evaluation Time Point
Description: The individual symptom score for Sneezing was rated on a 5-point
  scale of severity using the following scale: 0 = None (No symptoms), 1 = MILD (Symptom is present, but easily tolerated), 2 = MODERATE (Awareness of symptoms, bothersome, but tolerable), 3 = SEVERE (Definite awareness of symptoms, difficult to tolerate but does not interfere with activities), 4 = VERY SEVERE (Difficult to tolerate and interferes with the activities of daily living). The Sneezing symptom score ranges from 0 - 5. Increasing scores are associated with increasing severity.
Time Frame: From time of sensitization (time 0) to end of visit (~8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Loratadine | Fexofenadine | Placebo
Number analyzed (Participants) | 85 | 85 | 85
units on a scale
  0 minutes (n=85, n=85, n=85) | 1.3 (1.37) | 1.2 (1.36) | 1.5 (1.40)
  15 minutes (n=85, n=85, n=85) | 1.2 (1.31) | 1.2 (1.39) | 1.3 (1.37)
  30 minutes (n=85, n=85, n=85) | 1.2 (1.34) | 1.1 (1.32) | 1.2 (1.38)
  45 minutes (n=85, n=85, n=85) | 1.0 (1.29) | 0.9 (1.22) | 1.3 (1.39)
  60 minutes (n=85, n=85, n=85) | 1.1 (1.21) | 0.7 (1.12) | 1.2 (1.36)
  75 minutes (n=85, n=85, n=85) | 1.0 (1.25) | 0.8 (1.16) | 1.1 (1.39)
  90 minutes (n=85, n=85, n=85) | 0.7 (1.12) | 0.6 (1.07) | 1.0 (1.37)
  105 minutes (n=85, n=85, n=85) | 0.8 (1.16) | 0.6 (1.07) | 1.1 (1.43)
  120 minutes (n=85, n=85, n=85) | 0.5 (0.88) | 0.5 (1.04) | 0.9 (1.28)
  135 minutes (n=85, n=85, n=85) | 0.8 (1.13) | 0.7 (1.20) | 1.2 (1.48)
  150 minutes (n=85, n=85, n=85) | 0.9 (1.22) | 0.6 (1.14) | 1.1 (1.32)
  165 minutes (n=85, n=85, n=85) | 0.8 (1.11) | 0.5 (1.03) | 0.9 (1.32)
  180 minutes (n=85, n=85, n=85) | 0.7 (1.08) | 0.6 (1.11) | 0.9 (1.30)
  195 minutes (n=85, n=85, n=85) | 0.8 (1.19) | 0.6 (1.09) | 1.0 (1.38)
  210 minutes (n=85, n=85, n=85) | 0.7 (1.07) | 0.5 (1.03) | 1.0 (1.31)
  225 minutes (n=85, n=85, n=85) | 0.7 (1.04) | 0.6 (0.93) | 0.9 (1.33)
  240 minutes (n=85, n=85, n=85) | 0.7 (1.09) | 0.5 (1.04) | 0.9 (1.29)
  255 minutes (n=85, n=85, n=85) | 0.6 (1.15) | 0.4 (0.86) | 1.0 (1.41)
  270 minutes (n=85, n=85, n=85) | 0.6 (1.13) | 0.5 (1.00) | 1.0 (1.40)
  285 minutes (n=85, n=85, n=85) | 0.8 (1.08) | 0.6 (1.07) | 1.1 (1.42)
  300 minutes (n=84, n=85, n=85) | 0.7 (1.02) | 0.5 (0.95) | 0.9 (1.34)
  315 minutes (n=84, n=85, n=85) | 0.7 (1.10) | 0.4 (0.94) | 1.1 (1.40)
  330 minutes (n=85, n=85, n=85) | 0.7 (1.02) | 0.6 (1.03) | 1.0 (1.38)
  345 minutes (n=84, n=85, n=85) | 0.7 (1.09) | 0.6 (0.99) | 1.0 (1.33)
  360 minutes (n=85, n=85, n=85) | 0.6 (1.12) | 0.6 (1.09) | 1.0 (1.38)

5. Secondary Outcome: Mean Individual Symptom Scores for Watery Eyes by Post-Treatment Evaluation Time Point
Description: The individual symptom score for Water Eyes was rated on a 5-point
  scale of severity using the following scale: 0 = None (No symptoms), 1 = MILD (Symptom is present, but easily tolerated), 2 = MODERATE (Awareness of symptoms, bothersome, but tolerable), 3 = SEVERE (Definite awareness of symptoms, difficult to tolerate but does not interfere with activities), 4 = VERY SEVERE (Difficult to tolerate and interferes with the activities of daily living). The Watery Eyes symptom score ranges from 0 - 5. Increasing scores are associated with increasing severity.
Time Frame: From time of sensitization (time 0) to end of visit (~8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Loratadine | Fexofenadine | Placebo
Number analyzed (Participants) | 85 | 85 | 85
units on a scale
  0 minutes | 2.7 (1.12) | 2.8 (1.05) | 2.7 (1.02)
  15 minutes | 2.4 (1.17) | 2.6 (1.10) | 2.4 (1.15)
  30 minutes | 2.2 (1.23) | 2.3 (1.17) | 2.1 (1.25)
  45 minutes | 1.9 (1.22) | 2.0 (1.19) | 2.0 (1.18)
  60 minutes | 1.8 (1.21) | 1.9 (1.16) | 1.9 (1.12)
  75 minutes | 1.7 (1.21) | 1.8 (1.19) | 1.6 (1.11)
  90 minutes | 1.5 (1.29) | 1.6 (1.23) | 1.5 (1.18)
  105 minutes | 1.5 (1.22) | 1.6 (1.13) | 1.5 (1.19)
  120 minutes | 1.3 (1.15) | 1.3 (1.09) | 1.4 (1.18)
  135 minutes | 1.2 (1.11) | 1.3 (1.11) | 1.4 (1.29)
  150 minutes | 1.2 (1.12) | 1.2 (1.19) | 1.4 (1.20)
  165 minutes | 1.2 (1.14) | 1.2 (1.14) | 1.4 (1.20)
  180 minutes | 1.2 (1.07) | 1.1 (1.12) | 1.3 (1.16)
  195 minutes | 1.2 (1.15) | 1.2 (1.19) | 1.5 (1.21)
  210 minutes | 1.2 (1.14) | 1.1 (1.13) | 1.4 (1.27)
  225 minutes | 1.2 (1.13) | 1.1 (1.16) | 1.4 (1.25)
  240 minutes | 1.2 (1.16) | 1.1 (1.10) | 1.4 (1.24)
  255 minutes | 1.2 (1.12) | 1.1 (1.13) | 1.4 (1.26)
  270 minutes | 1.2 (1.13) | 1.1 (1.09) | 1.4 (1.21)
  285 minutes | 1.2 (1.08) | 1.2 (1.13) | 1.4 (1.27)
  300 minutes | 1.2 (1.02) | 1.1 (1.10) | 1.3 (1.32)
  315 minutes | 1.2 (1.09) | 1.2 (1.13) | 1.4 (1.33)
  330 minutes | 1.3 (1.14) | 1.2 (1.15) | 1.4 (1.32)
  345 minutes | 1.2 (1.15) | 1.2 (1.19) | 1.4 (1.32)
  360 minutes | 1.2 (1.20) | 1.3 (1.17) | 1.4 (1.34)

6. Secondary Outcome: Mean Individual Symptom Scores for Itchy Eyes by Post-Treatment Evaluation Time Point
Description: The individual symptom score for Itchy Eyes was rated on a 5-point
  scale of severity using the following scale: 0 = None (No symptoms), 1 = MILD (Symptom is present, but easily tolerated), 2 = MODERATE (Awareness of symptoms, bothersome, but tolerable), 3 = SEVERE (Definite awareness of symptoms, difficult to tolerate but does not interfere with activities), 4 = VERY SEVERE (Difficult to tolerate and interferes with the activities of daily living). The Itchy Eyes symptom score ranges from 0 - 5. Increasing scores are associated with increasing severity.
Time Frame: From time of sensitization (time 0) to end of visit (~8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Loratadine | Fexofenadine | Placebo
Number analyzed (Participants) | 85 | 85 | 85
units on a scale
  0 minutes (n=85, n=85, n=85) | 3.0 (0.93) | 3.2 (0.87) | 3.1 (1.08)
  15 minutes (n=85, n=85, n=84) | 2.6 (1.10) | 3.0 (1.02) | 2.8 (1.15)
  30 minutes (n=85, n=85, n=85) | 2.4 (1.12) | 2.7 (1.17) | 2.4 (1.20)
  45 minutes (n=85, n=85, n=85) | 2.2 (1.14) | 2.3 (1.17) | 2.4 (1.24)
  60 minutes (n=85, n=85, n=85) | 1.9 (1.14) | 2.1 (1.14) | 2.2 (1.23)
  75 minutes (n=85, n=85, n=85) | 1.9 (1.14) | 2.0 (1.20) | 1.9 (1.25)
  90 minutes (n=85, n=85, n=85) | 1.8 (1.21) | 1.8 (1.17) | 1.9 (1.28)
  105 minutes (n=85, n=85, n=85) | 1.8 (1.18) | 1.8 (1.15) | 1.8 (1.29)
  120 minutes (n=85, n=85, n=85) | 1.6 (1.19) | 1.6 (1.14) | 1.7 (1.30)
  135 minutes (n=85, n=85, n=85) | 1.5 (1.14) | 1.5 (1.13) | 1.7 (1.28)
  150 minutes (n=85, n=85, n=85) | 1.5 (1.06) | 1.4 (1.20) | 1.6 (1.32)
  165 minutes (n=85, n=85, n=85) | 1.5 (1.11) | 1.4 (1.24) | 1.7 (1.28)
  180 minutes (n=85, n=85, n=85) | 1.4 (1.11) | 1.4 (1.18) | 1.7 (1.23)
  195 minutes (n=85, n=85, n=85) | 1.5 (1.15) | 1.4 (1.19) | 1.8 (1.30)
  210 minutes (n=85, n=85, n=85) | 1.4 (1.12) | 1.4 (1.21) | 1.7 (1.26)
  225 minutes (n=85, n=85, n=85) | 1.5 (1.15) | 1.4 (1.19) | 1.7 (1.28)
  240 minutes (n=84, n=85, n=85) | 1.6 (1.19) | 1.4 (1.11) | 1.7 (1.29)
  255 minutes (n=85, n=85, n=85) | 1.4 (1.13) | 1.4 (1.18) | 1.6 (1.31)
  270 minutes (n=85, n=85, n=85) | 1.4 (1.09) | 1.4 (1.15) | 1.6 (1.30)
  285 minutes (n=85, n=85, n=85) | 1.3 (1.16) | 1.4 (1.17) | 1.7 (1.42)
  300 minutes (n=85, n=85, n=85) | 1.4 (1.19) | 1.4 (1.18) | 1.7 (1.33)
  315 minutes (n=85, n=85, n=85) | 1.4 (1.19) | 1.4 (1.24) | 1.7 (1.36)
  330 minutes (n=85, n=85, n=85) | 1.5 (1.21) | 1.4 (1.24) | 1.6 (1.38)
  345 minutes (n=85, n=85, n=85) | 1.4 (1.23) | 1.4 (1.27) | 1.8 (1.38)
  360 minutes (n=85, n=85, n=85) | 1.5 (1.34) | 1.4 (1.25) | 1.7 (1.37)

7. Secondary Outcome: Mean Individual Symptom Scores for Nasal Congestion by Post-Treatment Evaluation Time Point
Description: The individual symptom score for Nasal Congestion was rated on a 5-point
  scale of severity using the following scale: 0 = None (No symptoms), 1 = MILD (Symptom is present, but easily tolerated), 2 = MODERATE (Awareness of symptoms, bothersome, but tolerable), 3 = SEVERE (Definite awareness of symptoms, difficult to tolerate but does not interfere with activities), 4 = VERY SEVERE (Difficult to tolerate and interferes with the activities of daily living). The Nasal Congestion symptom score ranges from 0 - 5. Increasing scores are associated with increasing severity.
Time Frame: From time of sensitization (time 0) to end of visit (~8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Loratadine | Fexofenadine | Placebo
Number analyzed (Participants) | 85 | 85 | 85
units on a scale
  0 minutes (n=85, n=85, n=85) | 3.4 (0.81) | 3.2 (0.88) | 3.4 (0.76)
  15 minutes (n=85, n=85, n=85) | 2.5 (1.20) | 2.2 (1.25) | 2.7 (1.19)
  30 minutes (n=85, n=85, n=85) | 1.6 (1.33) | 1.5 (1.19) | 2.0 (1.26)
  45 minutes (n=85, n=85, n=85) | 2.5 (1.16) | 2.1 (1.21) | 2.6 (1.22)
  60 minutes (n=85, n=85, n=85) | 1.6 (1.29) | 1.4 (1.20) | 1.8 (1.34)
  75 minutes (n=85, n=85, n=85) | 2.4 (1.25) | 2.1 (1.21) | 2.6 (1.24)
  90 minutes (n=85, n=85, n=85) | 1.6 (1.27) | 1.3 (1.19) | 1.8 (1.34)
  105 minutes (n=85, n=85, n=85) | 2.4 (1.24) | 2.1 (1.20) | 2.6 (1.24)
  120 minutes (n=85, n=85, n=85) | 1.5 (1.26) | 1.4 (1.17) | 1.8 (1.31)
  135 minutes (n=85, n=85, n=85) | 2.4 (1.24) | 2.1 (1.19) | 2.6 (1.26)
  150 minutes (n=85, n=85, n=85) | 1.5 (1.31) | 1.3 (1.19) | 1.8 (1.31)
  165 minutes (n=85, n=85, n=85) | 2.4 (1.26) | 2.0 (1.14) | 2.5 (1.33)
  180 minutes (n=85, n=85, n=85) | 1.4 (1.22) | 1.3 (1.22) | 1.8 (1.39)
  195 minutes (n=85, n=85, n=85) | 2.5 (1.21) | 2.0 (1.15) | 2.6 (1.25)
  210 minutes (n=85, n=85, n=85) | 1.5 (1.31) | 1.3 (1.20) | 1.8 (1.34)
  225 minutes (n=85, n=85, n=85) | 2.4 (1.21) | 2.0 (1.24) | 2.6 (1.28)
  240 minutes (n=85, n=85, n=85) | 1.5 (1.29) | 1.4 (1.21) | 1.8 (1.32)
  255 minutes (n=85, n=85, n=84) | 2.4 (1.26) | 2.0 (1.19) | 2.6 (1.30)
  270 minutes (n=85, n=85, n=84) | 1.6 (1.29) | 1.3 (1.22) | 1.8 (1.46)
  285 minutes (n=85, n=85, n=85) | 2.4 (1.31) | 2.1 (1.19) | 2.6 (1.34)
  300 minutes (n=85, n=85, n=85) | 1.5 (1.31) | 1.3 (1.25) | 1.8 (1.43)
  315 minutes (n=85, n=85, n=85) | 2.4 (1.29) | 2.1 (1.19) | 2.5 (1.39)
  330 minutes (n=85, n=85, n=85) | 1.5 (1.31) | 1.3 (1.24) | 1.8 (1.47)
  345 minutes (n=85, n=85, n=85) | 2.4 (1.28) | 2.0 (1.24) | 2.5 (1.33)
  360 minutes (n=85, n=85, n=85) | 1.5 (1.31) | 1.4 (1.31) | 1.9 (1.51)

8. Secondary Outcome: Mean Individual Symptom Scores for Itchy Mouth/Throat/Ears by Post-Treatment Evaluation Time Point
Description: The individual symptom score for Itchy Mouth/Throat/Ears was rated on a 5-point
  scale of severity using the following scale: 0 = None (No symptoms), 1 = MILD (Symptom is present, but easily tolerated), 2 = MODERATE (Awareness of symptoms, bothersome, but tolerable), 3 = SEVERE (Definite awareness of symptoms, difficult to tolerate but does not interfere with activities), 4 = VERY SEVERE (Difficult to tolerate and interferes with the activities of daily living). The Itchy Mouth/Throat/Ears symptom score ranges from 0 - 5. Increasing scores are associated with increasing severity.
Time Frame: From time of sensitization (time 0) to end of visit (~8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Loratadine | Fexofenadine | Placebo
Number analyzed (Participants) | 85 | 85 | 85
units on a scale
  0 minutes (n=85, n=85, n=85) | 3.0 (1.08) | 3.0 (1.05) | 2.9 (1.17)
  15 minutes (n=85, n=85, n=85) | 3.2 (1.05) | 3.0 (1.06) | 3.0 (1.09)
  30 minutes (n=85, n=85, n=85) | 2.6 (1.19) | 2.8 (1.17) | 2.6 (1.27)
  45 minutes (n=85, n=85, n=85) | 3.0 (1.11) | 2.8 (1.09) | 2.8 (1.06)
  60 minutes (n=85, n=85, n=85) | 2.3 (1.29) | 2.6 (1.27) | 2.4 (1.25)
  75 minutes (n=85, n=85, n=85) | 2.8 (1.16) | 2.6 (1.16) | 2.8 (1.12)
  90 minutes (n=85, n=85, n=85) | 2.0 (1.22) | 2.3 (1.16) | 2.3 (1.25)
  105 minutes (n=85, n=85, n=85) | 2.7 (1.19) | 2.4 (1.17) | 2.6 (1.14)
  120 minutes (n=85, n=85, n=85) | 1.9 (1.24) | 2.0 (1.15) | 2.1 (1.31)
  135 minutes (n=85, n=85, n=85) | 2.6 (1.20) | 2.3 (1.24) | 2.5 (1.24)
  150 minutes (n=85, n=85, n=85) | 1.8 (1.21) | 1.8 (1.17) | 1.9 (1.32)
  165 minutes (n=85, n=85, n=85) | 2.5 (1.17) | 2.2 (1.21) | 2.4 (1.29)
  180 minutes (n=85, n=85, n=85) | 1.7 (1.20) | 1.7 (1.21) | 1.8 (1.29)
  195 minutes (n=85, n=85, n=85) | 2.4 (1.25) | 2.1 (1.17) | 2.4 (1.26)
  210 minutes (n=85, n=85, n=85) | 1.6 (1.21) | 1.7 (1.12) | 1.9 (1.28)
  225 minutes (n=85, n=85, n=85) | 2.3 (1.13) | 2.0 (1.20) | 2.3 (1.25)
  240 minutes (n=85, n=85, n=85) | 1.5 (1.18) | 1.5 (1.15) | 1.7 (1.31)
  255 minutes (n=85, n=85, n=84) | 2.3 (1.19) | 2.0 (1.22) | 2.4 (1.28)
  270 minutes (n=85, n=85, n=85) | 1.5 (1.20) | 1.6 (1.16) | 1.7 (1.29)
  285 minutes (n=85, n=85, n=85) | 2.4 (1.16) | 2.0 (1.26) | 2.4 (1.31)
  300 minutes (n=85, n=85, n=85) | 1.5 (1.14) | 1.4 (1.21) | 1.8 (1.32)
  315 minutes (n=85, n=85, n=85) | 2.4 (1.18) | 2.0 (1.23) | 2.4 (1.30)
  330 minutes (n=85, n=85, n=85) | 1.4 (1.19) | 1.4 (1.22) | 1.7 (1.23)
  345 minutes (n=85, n=85, n=85) | 2.3 (1.20) | 2.0 (1.25) | 2.5 (1.29)
  360 minutes (n=85, n=85, n=85) | 1.4 (1.17) | 1.3 (1.21) | 1.7 (1.27)

ADVERSE EVENTS:
Arm/Group | Loratadine | Fexofenadine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/85 | 0/85
Other Adverse Events (participants affected / at risk) | 0/85 | 0/85 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No